CLINICAL TRIAL: NCT06186492
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled, Safety, Tolerability, and Pharmacokinetic Study of Single Ascending Doses and Multiple Doses of WVE-006 in Healthy Participants
Brief Title: A Phase 1 Research Study to Evaluate Safety, Tolerability, and Pharmacokinetics of WVE-006 in Healthy Participants With Wild-type AAT Expression (RestorAATion-1)
Acronym: RestorAATion-1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wave Life Sciences Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: WVE-006-001
Record Dates: First submitted 2023-11-09; First posted 2024-01-02 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Alpha-1 Antitrypsin Deficiency
MeSH Terms: conditions — alpha 1-Antitrypsin Deficiency

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (7):
- Experimental WVE-006 (Dose A) or placebo (Experimental)
  Interventions: Drug: WVE-006
- Experimental WVE-006 (Dose B) or placebo (Experimental)
  Interventions: Drug: WVE-006
- Experimental WVE-006 (Dose C) or placebo (Experimental)
  Interventions: Drug: WVE-006
- Experimental WVE-006 (Dose D) or placebo (Experimental)
  Interventions: Drug: WVE-006
- Experimental WVE-006 (Dose E) or placebo (Experimental)
  Interventions: Drug: WVE-006
- Experimental WVE-006 (Dose F) or placebo (Experimental)
  Interventions: Drug: WVE-006
- Experimental WVE-006 (Dose G) or placebo (Experimental)
  Interventions: Drug: WVE-006

INTERVENTIONS:
Drug: WVE-006 — RNA editing oligonucleotide

SUMMARY:
This study is the first study in the RestorAATion clinical program.

The purpose of this first-in human (FIH), double-blind, randomized, placebo-controlled, single ascending dose (SAD) and multiple-dose Phase 1 study is to assess the safety, tolerability, and PK of WVE-006 compared to placebo in healthy participants following a single dose (Period 1) and multiple doses (Period 2) of WVE-006.

This information will be used to determine doses and regimes that have the potential to be pharmacologically active in patients with Alpha-1 antitrypsin deficiency in the RestorAATion 2 study, and the maximum safe and tolerable dose that may be given to these patients.

ELIGIBILITY:
Inclusion Criteria:

* Healthy as determined by the Investigator, based on a medical evaluation.
* Genetic testing confirming PI*MM.
* Participant has been a non-smoker for at least 1 year prior to screening.

Exclusion Criteria:

* Participant has a history of multiple drug allergies or of allergic reaction to an oligonucleotide or to N-acetylgalactosamine (GalNAc).
* Participant has a history of intolerance or any medical condition that might interfere with subcutaneous injections.
* Any ongoing or recent infections.
* Any recent or planned vaccinations during the study.
* Participant has a history of regular alcohol consumption exceeding 14 standard drinks/week.
* Unwilling to abstain from alcohol for 48 hours prior to dosing at each of the dosing visits.
* Participant has a history of caffeine consumption exceeding 8 cups of coffee/day.
* Use of prescription or non-prescription medications, including vitamin, dietary, and herbal supplements (including St John's Wort) within 7 days prior to the first dose of study treatment unless, in the opinion of the Investigator and Sponsor, the medication will not interfere with interpretation of study assessments. Contraception and hormone replacement therapy (HRT) are permitted. If needed, over-the-counter (OTC) medications such as paracetamol/acetaminophen may be used acutely.
* Any recent or planned major surgery during the study.
* Donation of blood or blood products in excess of 500 mL within 12 weeks prior to Screening Visit and/or unwilling to refrain from blood donation for the duration of the study.
* Participant has received an investigational agent within 3 months of the Screening Visit.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2023-11-14 (Actual); Primary Completion 2025-02-13 (Actual); Study Completion 2025-02-13 (Actual)

PRIMARY OUTCOMES:
The proportion of participants with adverse events | Day 1 through Day 85 after last dose.

SECONDARY OUTCOMES:
Single Ascending Dose - Area under the plasma concentration time curve for WVE-006 from time of dosing to the last measurable concentration (AUClast) | Day 0 through Day 84 postdose
Single Ascending Dose - Maximum concentration of WVE-006 in plasma (Cmax) | Day 0 through Day 84 postdose
Multiple Ascending Doses - Area under the plasma concentration time curve for WVE-006 from time of dosing to the last measurable concentration (AUClast) | Day 0-14 after the first and Day 0-84 days after the last dose, respectively
Multiple Ascending Doses - Maximum concentration of WVE-006 in plasma (Cmax) | Day 0-14 after the first and Day 0-84 days after the last dose, respectively

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Caracta, MD, Study Director — Wave Life Sciences
Locations (1):
- Simbec-Orion Clinical Pharmacology,, Merthyr Tydfil, Wales, United Kingdom

IPD SHARING:
Plan to Share IPD: No